CLINICAL TRIAL: NCT03022344
Title: Coronary Plaque Morphology and Plaque Progression in Patients With Newly Diagnosed Type-2 Diabetes Mellitus
Brief Title: DD2-Coronary Plaque Morphology and Plaque Progression
Acronym: DD2plaque
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: The Danish Diabetes Academy supported by the Novo Nordisk Foundation (Unknown); University of Southern Denmark (Other); Department of Regional Health Research - Center Southwest (Unknown); Edith and Vagn Hedegaard Jensens Foundation (Unknown); Karola Jørgensens Foundation and Foundation for Cardiology in Southwest Denmark. (Unknown)
Responsible Party: Principal Investigator, Monija Mrgan, MD, Esbjerg Hospital - University Hospital of Southern Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 44110
Record Dates: First submitted 2017-01-09; First posted 2017-01-16 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Diabetes; Plaque; Atherosclerosis
Keywords: DD2 plaque study; Coronary plaque; Type-2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus; Plaque, Amyloid; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy (Sham Comparator): Patients in this cohort consist of 100 healthy patients
  Interventions: Radiation: Cardiac CT
- Diabetes mellitus (Sham Comparator): Newly diagnosed (< 1 year) diabetes patients clinically classified as type-2 diabetes patients of both sex
  Interventions: Radiation: Cardiac CT

INTERVENTIONS:
Radiation: Cardiac CT

SUMMARY:
However, there is only very sparse information regarding the atherosclerotic burden and cardiovascular biomarkers in the early stages of type-2 diabetes, as the vast majority of studies have concerned diabetes populations with more than 5 years average diabetes age or high-risk subgroups, who at inclusion already had atherosclerotic disease manifestations.

Consequently, this study aims on evaluating the occurrence of early-stage subclinical atherosclerosis in newly diagnosed type-2 diabetes with special emphasis on coronary plaque characteristics by modern imaging techniques. These findings will be compared to the functional status of various peripheral arterial segments and biomarkers in the cross-sectional part of this study. The 5-year follow-up study intends to describe relationships between these selected measures for general atherosclerotic involvement and the progression of the coronary atherosclerotic burden by contemporary techniques.

DETAILED DESCRIPTION:
THE AIM

The objective of this study is to:

Study I: Compare the prevalence and complexity of coronary plaques in patients with newly discovered type-2 diabetes with a healthy control group matched for age and gender, as evaluated by coronary computed tomography angiography.

Study II: Describe the relationship between morphological, functional and biochemical estimates of arteriosclerosis in newly diagnosed type-2 diabetes.

Study III: Characterize the progression of coronary plaques in patients with newly discovered type-2 diabetes in a 5-year follow-up study.

DESIGN

"Coronary plaque morphology and plaque progression in patients with newly diagnosed type-2 diabetes mellitus" (DD2-plaque study) is a prospective cohort follow up study.

The inclusion phase will run for 2 years. The follow-up phase is 5 years from inclusion.

The DD2-plaque study (diabetic patient's cohort):

Recruitment in this cohort will take place in three ways:

1. From the "Danish centers for strategic research in type 2 diabetes" (DD2) - patients who agreed to be contacted for participation in a future study.
2. Direct from outpatient clinics in The Region of Southern. Patients will either be recruited through general practitioners or from outpatient clinics in The Region of Southern Denmark. The investigators expect to be able to include 100 asymptomatic patients with newly diagnosed type-2 diabetes.

Inclusion criteria

1. Newly diagnosed (< 1 year) diabetes patients clinically classified as type-2 diabetes patients of both sex.
2. Age 18 +.

Exclusion criteria

1. Type 1 diabetes (or have age<30 years and C-peptid<300pmol/l and GAD-ab titer> 20 IU/ml).
2. Renal insufficiency (GFR < 45 or se-creatinine >140 micromol/l).
3. BMI > 35 kg/m2
4. Atrial fibrillation.
5. Life expectancy below 2 years.
6. Mental disease and/or misuse of alcohol or drugs that affects patient's ability to give informed consent.
7. Pregnancy at time of or planned at inclusion.
8. Patients with a history of prior atherothrombotic disease (including acute coronary syndromes, prior revascularization, ischemic stroke or peripheral arterial disease).

The DD2-plaque study (control patients cohort):

100 controls will be recruited from the general population by advertisement in the local press. Controls with cardiovascular disease (criteria consistent with those described for patients with type-2 diabetes) and type-2 diabetes (undiagnosed type-2 diabetes in this group was excluded by fasting plasma glucose and by an oral glucose tolerance test) will be excluded. In addition, exclusion criteria are also consistent with those described for patients with type-2 diabetes.

Longitudinal measurements will be done at the screening visit and after 5 years.

1. The proxy statement.
2. Participants will fill in a questionnaire concerning:

   * Cardiovascular and diabetes hereditary
   * Medication
   * Alcohol and drugs consumption
   * Smoking habits (current, prior and never smokers)
   * Family history (cardiac events or strokes for women < 65 years of age and men < 55 years of age in first generation relatives)
   * Medical history
3. Physical examination will include measurement of:

   * Height, weight, BMI.
   * Waist/hip ratio
   * ECG
4. Brachial blood pressure will be measured by oscillometric technics during 24 hours using TM-2430 (A&D CO., LTD, Saitama, Japan) or BDM Mobil-O-Graph® NG Classic (IEM GmbH, Stolberg, Germany).
5. Blood samples: Procedures for handling and shipping samples is available in the trial master and at www.DD2.nu under "blodprøvetagning".

   An exception to these procedures are that the blood samples will be frozen at site and send on ice to the biobank.

   2 x 9 ml. containers with green lid (Li-hep) 2 x 2.7 ml. containers with blue lid (Na-citrat) 2 x 9 ml. containers with purple lid (EDTA) 2 x 4 ml. containers with purple/dark purple lid (EDTA) 2 x 3 ml. containers with pink lid (Fluoridcitrat) 2 x 9 ml. containers with brown lid (Serum)

   1 container for urine with yellow lid 10 ml of morning midstream urine will be sampled. Urine sticks will be used to rule out urinary tract infection. If this is present the urine should be resembled. A total of 73.4 ml + 10 ml of blood will be drawn.

   For a subset of patients the DD2 cohort registration and the baseline visit will take place in the same day. These patients will have 146.8 ml of blood drawn on the same day. Containers will be sent to the patients.
6. Biochemical analysis: total cholesterol, S-LDL-cholesterol, S-HDL-cholesterol and S-triglycerides, HbA1c, glucose, C-reactive protein, D-dimer, creatinin and fibrinogen. All analyses are performed at our local Dept. of Clinical Biochemistry.
7. All patients will undergone:

   Carotid intima media thickness (IMT) will be measured by B-mode ultrasound (Model IE33, Koninklijke Philips Electronics N.V, Eindhoven, The Netherlands) using a linear array transducer, L11-3 with a frequency up to 11 MHz.
8. Pulse wave velocity: Using sphygmocor (ArtCor, Sydney, Australia).
9. Ankle brachial index.
10. Albumin creatinine ratio
11. Coronary atherosclerosis is evaluated by measurement of calcium in the coronary arteries and by evaluation of coronary plaques using contrast enhanced cardiac CT. Coronary artery calcifications will be estimated by the Agatston score while the evaluation of coronary plaques will be performed by a dedicated plaque-analysis tool, Auto-Plaque.

STATISTICS

Sample size estimations are performed for comparison of calcium scoring between patients with type-2 diabetes and normal controls (Un-paired evaluation) and comparison of calcium scoring between type-2 diabetes patients at inclusion and at follow-up (Paired). From previous studies on calcium scoring in the Danish Risk Score Study cohort, the standard deviation, SD, on coronary calcification is known to be 32.7 UE (Agatston Score). It is supposed that SD in the diabetic patients is equal to the figure in controls. Under the assumptions that 15% will drop-out, a MIREDIF of 20 (twice the threshold for registering the occurrence of coronary calcification in the central West Danish Heart Registry, VDH), beta= 0, 1 and alfa= 0.02 (Planned comparative analysis of 2-3 plaque-components) it is calculated, that it is needed to include 41 patients in each group for the un-paired analyses and to follow 41 diabetic patients for 5 years (Paired analysis). It is supposed, that app. 40% of type-2 diabetes patients meet the age criteria (55+/-5 years or 65+/-5 years) for comparison with the background population, which means that app. 100 type-2 diabetes patients should be included in the DD2 plaque study.

Students T-test will be used for comparison of normally distributed continuous variables and the Mann-Whitney test will be used for comparison of continuous variables that are not normally distributed. The χ2- test is performed for comparison of dichotomous variables. Continuous variables are presented as either mean or standard deviation or median and interquartile range. P-values <0.05 will be considered statistically significant. Stepwise multivariate logistic regression will be performed for analysis of which factors are associated with coronary atherosclerosis using either presence coronary artery calcification or other plaque variables as dependant variables.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed (< 1 year) diabetes patients clinically classified as type-2 diabetes patients of both sex.
* Age 18 +.

Exclusion Criteria:

* Type 1 diabetes (or have age<30 years and C-peptid<300pmol/l and GAD-ab titer> 20 IU/ml).
* Renal insufficiency (GFR < 45 or se-creatinine >140 micromol/l).
* BMI > 35.
* Atrial fibrillation.
* Life expectancy below 2 years.
* Mental disease and/or misuse of alcohol or drugs that affects patient's ability to give informed consent.
* Pregnancy at time of or planned at inclusion.
* Patients with a history of prior atherothrombotic disease (including acute coronary syndromes, prior revascularization, ischemic stroke or peripheral arterial disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-11; Primary Completion 2021-06 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Progression of contrast enhanced cardiac CT in relation to baseline and follow-up cardiovascular risk factors and biomarkers. | 5 years
  Coronary artery calcification were quantified by non-contrast cardiac CT and were assessed by summing up the scores from all foci in the coronary arteries, expressed in Agatston units (U), using dedicated software (Syngo Calcium scoring, (Siemens Healthcare).

SECONDARY OUTCOMES:
Biochemical analysis in relation to contrast enhanced cardiac CT | 1 year
  no. of participants with abnormal laboratory values compared to abnormal/normal enhanced cardiac CT
Body mass index (kg/m2) | 1 year
  Cardiovascular risk factors. No of participants with body mass index > 30 kg/m2
Carotid intima media thickness | 1 year
  A measure of the combined thickness of intima and media layers of carotid artery, assessed by B-mode ultrasound.values between 0.6 and 0.7 mm have been considered normal. Values > 1 mm or more has been associated with significant increased absolute risk of atherosclerosis. No of participants with values > 1 mm.
Ankle brachial index | 1year
  An ankle brachial index between and including 0.9 and 1.2 considered normal (free from significant peripheral artery disease), while a lesser than 0.9 indicates arterial disease. No of participants with value < 0.9.
waist hip ratio (m) | 1 year
  Abdominal obesity was defined as a waist-hip ratioabove 0.90 for males and above 0.85 for females,or a body mass index above 30.0 kg/m2. No of participants with abdominal obesity
Blood pressure (mmHg) | 1 year
  Hypertension was defined as blood pressures ≥ 140/90. No of participants with hypertension

CONTACTS AND LOCATIONS:
Locations (1):
- Sydvestjysk sygehus, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: No